CLINICAL TRIAL: NCT05417308
Title: A Pilot Trial of Topical vs Oral Minoxidil for Treatment of Endocrine Therapy-Induced Alopecia in Breast Cancer Patients
Brief Title: Topical or Oral Minoxidil for the Treatment of Endocrine Therapy-Induced Alopecia in Patients With Stage I-IV Breast Cancer
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ohio State University Comprehensive Cancer Center (Other)
Responsible Party: Principal Investigator, Brittany Dulmage, Principal Investigator, Ohio State University Comprehensive Cancer Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OSU-20340; NCI-2021-01932 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-03-16; First posted 2022-06-14 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-03

CONDITIONS: Anatomic Stage I Breast Cancer AJCC v8; Anatomic Stage IA Breast Cancer AJCC v8; Anatomic Stage IB Breast Cancer AJCC v8; Anatomic Stage II Breast Cancer AJCC v8; Anatomic Stage IIA Breast Cancer AJCC v8; Anatomic Stage IIB Breast Cancer AJCC v8; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IIIA Breast Cancer AJCC v8; Anatomic Stage IIIB Breast Cancer AJCC v8; Anatomic Stage IIIC Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Endocrine Therapy-Induced Alopecia; Prognostic Stage I Breast Cancer AJCC v8; Prognostic Stage IA Breast Cancer AJCC v8; Prognostic Stage IB Breast Cancer AJCC v8; Prognostic Stage II Breast Cancer AJCC v8; Prognostic Stage IIA Breast Cancer AJCC v8; Prognostic Stage IIB Breast Cancer AJCC v8; Prognostic Stage III Breast Cancer AJCC v8; Prognostic Stage IIIA Breast Cancer AJCC v8; Prognostic Stage IIIB Breast Cancer AJCC v8; Prognostic Stage IIIC Breast Cancer AJCC v8; Prognostic Stage IV Breast Cancer AJCC v8
MeSH Terms: interventions — Minoxidil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm I (topical minoxidil) (Active Comparator): Patients apply minoxidil foam topically to affected areas of the scalp QD for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Minoxidil; Other: Quality-of-Life Assessment; Other: Questionnaire Administration
- Arm II (orally minoxidil) (Experimental): Patients receive minoxidil PO QD for up to 12 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Minoxidil; Other: Quality-of-Life Assessment; Other: Questionnaire Administration

INTERVENTIONS:
Drug: Minoxidil — Applied topically
  Other Names: Alostil; Loniten; Rogaine; U 10858
  Arms: Arm I (topical minoxidil)
Drug: Minoxidil — Given PO
  Other Names: Alostil; Loniten; Rogaine; U 10858
  Arms: Arm II (orally minoxidil)
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This early phase I trial studies the possible benefits and/or side effects of topical or oral minoxidil in treating endocrine therapy-induced hair loss (alopecia) in patients with stage I-IV breast cancer. Endocrine therapy-induced alopecia (EIA) is a distressing side effect that leads to reduced quality of life and early cessation of therapy in women undergoing treatment for breast cancer. Patients on endocrine therapy commonly report hair loss or thinning. Minoxidil is a drug that may promote hair growth and reduce hair loss. Oral minoxidil may increase hair density in women with EIA, and work the same as topical minoxidil in treating EIA in patients with breast cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the safety and tolerability of low-dose oral minoxidil in patients with breast cancer and EIA.

II. To obtain preliminary data to support whether low-dose oral minoxidil is a reasonable alternative to topical minoxidil in patients with EIA.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM I: Patients apply minoxidil foam topically to affected areas of the scalp once daily (QD) for up to 12 months in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive minoxidil orally (PO) QD for up to 12 months in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Women >= 18 years of age
* Established diagnosis of breast cancer stages I-IV
* On endocrine therapy including tamoxifen or aromatase inhibitors with or without concurrent use of ovarian function suppression
* Self-reporting hair loss since starting endocrine therapy

Exclusion Criteria:

* Pregnant or nursing women
* Current chemotherapy use or prior chemotherapy use within the last 2 years
* History of scarring/cicatricial alopecia or alopecia areata
* Prior use of oral or topical minoxidil
* Prior or ongoing use of spironolactone
* Known sensitivity to minoxidil
* Untreated hypothyroidism or iron deficiency as determined by thyroid stimulating hormone (TSH) with reflex free T4 and ferritin level > 40 to be checked at the time of enrolling if not completed in the 12 months prior

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of days assigned medication was taken/applied | Up to 12 months
  For the oral minoxidil group, the proportion of pills taken will be reported with a 95% confidence interval. For the topical minoxidil group, the proportions of days medication was applied will be reported with a 95% confidence interval.

SECONDARY OUTCOMES:
Occurrence of at least one adverse event (AE) of grade 1 or higher | Up to 12 months
  Adverse events will be summarized using National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 with reporting of the number and percentage of patients affected. The total number of participants with AEs of any grade, and the total number of participants with grade 3 or higher AEs will be compared between randomized groups using Fisher's exact test.
Change in hair density | Baseline to 3 months
  At least mild-to-moderate improvement in hair density from baseline to 3 months as determined by a board-certified dermatologist from photographs. Will construct two-sided 95% confidence intervals for improvements from baseline and differences between randomized groups. Response will be dichotomized as no improvement versus moderate-to-significant improvement.
Change in hair density | Baseline to 6 months
  At least mild-to-moderate improvement in hair density from baseline to 6 months as determined by a board-certified dermatologist from photographs. Will construct two-sided 95% confidence intervals for improvements from baseline and differences between randomized groups. Response will be dichotomized as no improvement versus moderate-to-significant improvement.
Change in hair density | Baseline to 12 months
  At least mild-to-moderate improvement in hair density from baseline to 12 months as determined by a board-certified dermatologist from photographs. Will construct two-sided 95% confidence intervals for improvements from baseline and differences between randomized groups. Response will be dichotomized as no improvement versus moderate-to-significant improvement.
Chemotherapy Alopecia Distress Scale (CADS) score | At 3 months
  Patients will complete a a self-administered 17-item questionnaire
CADS score physical | At 6 months
  a self-administered 17-item questionnaire which categorizes questions into 4 subscales including physical
CADS score physical | At 6 months
  a self-administered 17-item questionnaire which categorizes questions into 4 subscales including physical relationship
CADS score emotional | At 12 months
  a self-administered 17-item questionnaire which categorizes questions into 4 subscales including emotional relationship
Patient-reported outcomes | At 3 months
  Mean responses to the symptom experience diary questions and the satisfaction items will be compared between groups via t-test.
Patient-reported outcomes | At 6 months
  Mean responses to the symptom experience diary questions and the satisfaction items will be compared between groups via t-test.
Patient-reported outcomes | At 12 months
  Mean responses to the symptom experience diary questions and the satisfaction items will be compared between groups via t-test.

CONTACTS AND LOCATIONS:
Overall Officials: Brittany L Dulmage, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (1):
- Ohio State University Comprehensive Cancer Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu